CLINICAL TRIAL: NCT01061983
Title: Electrical Stimulation of the Internal Capsule for Intractable OCD
Brief Title: Electrical Stimulation of the Internal Capsule for Intractable Obsessive-compulsive Disorder (OCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Benjamin Greenberg, Chief of Outpatient Services, Associate Professor of Psychiatry, Butler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000204
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep brain stimulation; Treatment refractory; Ventral internal capsule/ventral striatum; Neurosurgery; Neuroimaging
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Participants will receive deep brain stimulation.
  Interventions: Device: Medtronic Activa Deep Brain Stimulation

INTERVENTIONS:
Device: Medtronic Activa Deep Brain Stimulation — In DBS, thin wires are used to carry electric current to the parts of the brain involved in OCD symptoms. These wires are implanted surgically and are attached to battery operated stimulators usually implanted in the chest. The study doctor will adjust the settings of the electrical stimulation to optimize treatment for each participant.
  Other Names: Deep Brain Stimulation (DBS); Activa System; Medtronic Activa Deep Brain Stimulation Therapy System

SUMMARY:
This study will evaluate the safety and effectiveness of deep brain stimulation in treating people with severe and otherwise treatment-resistant obsessive-compulsive disorder. We also expect to determine how DBS affects brain activity in brain circuits strongly implicated in OCD, and how such effects may relate to symptom change. This treatment study therefore also permits a unique and crucial test of current neuroanatomical models of both OCD pathogenesis and mechanisms underlying the response to treatment.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a chronic and debilitating illness that affects between 2% and 3% of the adult population of the United States. People with OCD often experience persistent unwanted thoughts and carry out ritual-like behaviors to rid themselves of these obsessive thoughts. Additionally, OCD symptoms are usually tied with feelings of intense anxiety and functional impairment, making it important for people with OCD to seek effective treatment. Although there are currently many treatment options for OCD, including psychotherapy and medications such as serotonin reuptake inhibitors, between 40% and 60%of people with OCD only partially respond, or do not respond at all, to these treatment methods. Given the large percentage of people who do not respond to aggressive conventional treatments, alternative options are necessary for people with treatment-resistant OCD. Deep brain stimulation (DBS) is a procedure that involves the se of thin wires to carry electric current to parts of the brain associated with producing OCD symptoms. DBS has been effectively and safely used to treat movement disorders, such as Parkinson's disease, and may be beneficial in reducing OCD symptom severity. This study will evaluate the safety and efficacy of DBS in treating people with severe and treatment-resistant OCD.

Study participation through follow-up will last up to 2 years. Participants will be allowed to remain on any pre-surgical medications or behavioral therapy programs throughout the study. Before surgery, all participants will undergo a series of initial tests and examinations that will include psychiatric, medical, and neuropsychological histories and examinations.

Implantation of the devices will be performed at a single session. The leads that are inserted into the anterior limb of each internal capsule, will be implanted under local anesthesia. On the day of the surgery, participants will have a metal frame fixed to their heads for support during surgery, and magnetic resonance imagining (MRI) will be used to determine the exact placement of the wires. An extension wire will pass from the scalp area to the subclavicular region and connect each electrode to a subcutaneous implanted pulse generator (IPG), which will be implanted under general anesthesia. After placement of the DBS system, the patient will be admitted to the hospital for overnight observation for possible complications. Postoperative evaluation will consist of physical and neurological examinations, postoperative CBC, electrolyte panel, x-rays of the head, neck, and chest, a standard shunt series to ensure the integrity of connections, and a head CT scan to monitor for possible postoperative intracranial hemorrhage.

Surgical implantation will be followed by a three-week period with no stimulation, and then an intensive five-day preliminary outpatient stimulation trial, followed by longer-term outpatient stimulation. All patients will follow the same sequence of test conditions. The initial DBS testing will be open, followed by three blocks of testing in which the patients and investigators administering rating scales will not be informed of the stimulation condition. These three blocks will in general be three months long, but may be longer or shorter depending on the stability of any clinical improvement, and the possible emergence of symptom worsening. The remainder of the the study, up to the two-year study endpoint, will consist of a continuation phase of active open stimulation.

ELIGIBILITY:
Inclusion Criteria:

* OCD, diagnosed by Structural Clinical Interview for DSM-IV (SCID-IV), judged to be of disabling severity with a Yale-Brown Obsessive-Compulsive Scale (YBOCS) score of 28 and a Global Assessment of Function (GAF) score of 45 or less.
* Persistence of this level of impairment for a minimum of five years despite adequate trials of or intolerance to 3 or 4 selective serotonin transporter inhibitors including fluoxetine, sertraline, fluvoxamine, paroxetine and clomipramine alone and in combination with behavior therapy, and augmentation of one of the selective SRIs with clomipramine, a neuroleptic, and clonazepam.
* Age of at least eighteen years, and no more than 55 years.
* Able to understand and comply with instructions.
* Written informed consent.
* Either drug free or on a stable drug regime for at least 6 weeks.
* Good general health.

Exclusion Criteria:

* Current or past psychotic disorder.
* Any clinically significant neurological disorder or medical illness affecting brain function, other than motor tics or Gilles de la Tourette syndrome.
* Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI).
* Any surgical contraindications to undergoing DBS, including labeled contraindications for DBS and/or inability to undergo presurgical MRI (cardiac pacemaker, pregnancy, metal in body, severe claustrophobia), infection, coagulopathy, inability to undergo awake operation, significant cardiac or other medical risk factors for surgery.
* Current or unstably remitted substance abuse disorder.
* Pregnancy and women of childbearing age not using effective contraception.
* History of body dysmorphic disorder.
* History of severe personality disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2001-01; Primary Completion 2004-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Obsessive-compulsive disorder (OCD) severity (Yale-Brown Obsessive-Compulsive Scale) | Measured at baseline, then monthly for nine months, then every three months during the open continuation phase

SECONDARY OUTCOMES:
Depression severity (Hamilton Depression Scale), Anxiety (Hamilton Anxiety Scale), and neuropsychological battery. | At baseline, monthly for 9 months, then every 3 months for the continuation of the open phase.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Greenberg, MD, PhD, Principal Investigator — Butler Hospital/Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Greenberg BD, Gabriels LA, Malone DA Jr, Rezai AR, Friehs GM, Okun MS, Shapira NA, Foote KD, Cosyns PR, Kubu CS, Malloy PF, Salloway SP, Giftakis JE, Rise MT, Machado AG, Baker KB, Stypulkowski PH, Goodman WK, Rasmussen SA, Nuttin BJ. Deep brain stimulation of the ventral internal capsule/ventral striatum for obsessive-compulsive disorder: worldwide experience. Mol Psychiatry. 2010 Jan;15(1):64-79. doi: 10.1038/mp.2008.55. Epub 2008 May 20. PMID 18490925
- [Result] Greenberg BD, Malone DA, Friehs GM, Rezai AR, Kubu CS, Malloy PF, Salloway SP, Okun MS, Goodman WK, Rasmussen SA. Three-year outcomes in deep brain stimulation for highly resistant obsessive-compulsive disorder. Neuropsychopharmacology. 2006 Nov;31(11):2384-93. doi: 10.1038/sj.npp.1301165. Epub 2006 Jul 19. PMID 16855529
- [Result] Rauch SL, Dougherty DD, Malone D, Rezai A, Friehs G, Fischman AJ, Alpert NM, Haber SN, Stypulkowski PH, Rise MT, Rasmussen SA, Greenberg BD. A functional neuroimaging investigation of deep brain stimulation in patients with obsessive-compulsive disorder. J Neurosurg. 2006 Apr;104(4):558-65. doi: 10.3171/jns.2006.104.4.558. PMID 16619660